CLINICAL TRIAL: NCT04428918
Title: Biospecimen Procurement for Immunological Landscape Studies Following Hematopoietic Cell Transplantation
Status: Withdrawn | Type: Observational
Why Stopped: The study was closed due to investigator discretion based on the lack of ability to recruit patients and research goals of the program.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200072; 20-C-0072
Record Dates: First submitted 2020-06-11; First posted 2020-06-11 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cell Transplantation; Hematologic Malignancies
Keywords: Immunological; Apheresis Products; Protein
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Allogeneic HCT recipient or patient pending receipt of HCT

SUMMARY:
Background:

Allogenic hematopoietic cell transplantation (HCT) is a procedure in which a person gets stem cells from a donor in order to treat their disease. Researchers want to collect samples from people who have had or will have HCT. They will perform tests on the samples to study the immune system and its response to infections and disease.

Objective:

To collect biological samples from people who have had or are planning to have HCT to treat primary immunodeficiencies, blood cancers, or disorders of T-cell proliferation and/or dysregulation.

Eligibility:

People age 8 years and older who have undergone or are planning to undergo HCT.

Design:

Participants will be screened with:

Medical history

Medical chart review

Physical exam

Blood tests.

Participants may give blood and urine samples.

Participants may have a skin biopsy.

Participants may undergo apheresis. For this, a needle will be placed into an arm vein to take blood. A machine divides the whole blood into parts. The sample cells are taken out and the rest of the blood is returned through a second needle in the other arm.

Participants may have a bone marrow aspiration and biopsy. For this, the hipbone will be numbed. A needle will be put into the hipbone. Bone marrow will be taken out through the needle.

Participants may have a tumor or other abnormal tissue biopsy. For this, a tissue sample is obtained using a needle and syringe. They will sign a separate consent form. They may have a body scan or ultrasound to help locate the tumor during the biopsy.

Participation lasts for as long as participants choose to give samples.

DETAILED DESCRIPTION:
Background:

* Allogenic Hematopoietic Cell Transplantation (HCT) is a potentially curative option for some patients with primary immunodeficiencies (PID) and hematological cancers.
* HCT for PID looks to restore defects in cells of hematopoietic origin allowing for eradication of protracted or recurrent viral infections.
* The curative potential of allogenic HCT for hematologic malignancies is mediated by the allogeneic immune system through a graft-versus-tumor (GVT) effect.
* Characterization of the immunologic landscape in patients with successful eradication of viral infections and hematologic malignancies following allogenic HCT requires further investigation.

Objectives:

-To collect and bank blood, apheresis products, tumor, body fluids, and other biospecimens from patients with allogenic HCT and perform immunological landscape studies.

Eligibility:

-Patients age greater than or equal to 8 years of age and have undergone or are planning to undergo HCT.

Design:

* Up to 100 subjects will be enrolled.
* Patients may undergo sampling of blood, apheresis products, tumor, effusions, ascites, urine, bone marrow, skin, mucosa, saliva, stool, sputum, spinal fluid, or other tissues or fluids for banking and laboratory studies.
* No investigational or experimental therapy will be given as part of this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of a hematologic malignancy, immunodeficiency or disorder of T-cell proliferation and/or dysregulation
* Have undergone or planning to undergo an allogenic hematopoietic cell transplantation
* Age greater than or equal to 8 years
* Additional inclusion criteria pertinent only for patients undergoing apheresis
* Hemoglobin greater than or equal to 8 mg/dL and platelet count > 75 K/uL
* Weight greater than or equal to 48 kg
* Adequate venous access

EXCLUSION CRITERIA:

* Active concomitant medical or psychological illnesses that may increase the risk to the subject
* Inability of subject or parent/legal guardian to provide informed consent
* Pregnant or breastfeeding women as some tests and procedures allowed are contraindicated in pregnancy (i.e., CT scans, administration of iodinated contrast)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients age > 8 years of age and have undergone or are planning to undergo HCT. Participants are selected from other NIH protocols (including screening protocols) they may be co-enrolled on and can include both inpatient and outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Sample Aquisition | Ongoing
  To conduct immunological landscape studies on samples collected. To collect and bank blood, apheresis products, tumor, body fluids, and other biospecimens from patients with allogenic HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0072.html